CLINICAL TRIAL: NCT04009200
Title: The Effect of Preoperative Anxiety on Postoperative Delirium in Children Who Will Undergo Circumcision Surgery
Brief Title: The Effect of Preoperative Anxiety on Postoperative Delirium in Children
Status: Completed | Type: Observational
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkay baran akkuş, specialist doctor, Ankara Diskapi Training and Research Hospital
Other Study IDs: 44/07
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Preoperative Anxiety; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- circumcision: Modified Yale Preoperative Anxiety Scores (m-YPAS), Visual Analogue Scale Anxiety (VAS-anxiety) will be evaluated when patients are taken to the preoperative waiting room.
  After awakening, patients will be taken to the postoperative wake-up room where Pediatric Anesthesia Recovery Delirium Scores (PAED), Recovery Agitation 5-point Scores (EA), FLACC scores will be evaluated every 5 minutes and mean arterial pressure, pulse, SPO2 values will be recorded. Duration of stay in recovery unit will be recorded
- inguinal hernia: Modified Yale Preoperative Anxiety Scores (m-YPAS), Visual Analogue Scale Anxiety (VAS-anxiety) will be evaluated when patients are taken to the preoperative waiting room.
  After awakening, patients will be taken to the postoperative wake-up room where Pediatric Anesthesia Recovery Delirium Scores (PAED), Recovery Agitation 5-point Scores (EA), FLACC scores will be evaluated every 5 minutes and mean arterial pressure, pulse, SPO2 values will be recorded. Duration of stay in recovery unit will be recorded

SUMMARY:
Investigation of the effect of preoperative anxiety on postoperative delirium in children who will undergo circumcision operation

DETAILED DESCRIPTION:
In order to determine the effect of circumcision on preoperative anxiety and postoperative delirium, patients will be divided into two groups who will undergo circumcision surgery and who will undergo inguinal hernia surgery.

Modified Yale Preoperative Anxiety Scores (m-YPAS), Visual Analogue Scale Anxiety (VAS-anxiety) will be evaluated when patients are taken to the preoperative waiting room.

After awakening, patients will be taken to the postoperative wake-up room where Pediatric Anesthesia Recovery Delirium Scores (PAED), Recovery Agitation 5-point Scores (EA), FLACC scores will be evaluated every 5 minutes and mean arterial pressure, pulse, SPO2 values will be recorded. Duration of stay in recovery unit will be recorded

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Elective circumcision or elective inguinal hernia

Exclusion Criteria:

* Chronic diseases
* Development disability
* Prematurity
* Neurological diseases
* Psychoactive medication use
* Hearing/ visual impairment
* History of surgery

Ages: 6 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — circumcision surgery is applied only to male patients
Study Population: First 60 patients coming to the operating room who met the study criteria
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety difference between groups | Before premedication, in operating room
  Preoperative anxiety will be evaluated by mYPAS (modified Yale Preoperative Anxiety Scale). The mYPAS consists of 22 items in five categories (activity, emotional expressivity, state of arousal, vocalization and use of parents). The highest behavioral level observed in each of the five mYPAS categories is the score for that category. Partial weights were calculated and then added to a total score that ranged from 0 to 100. Cut off points were set to classify: a score of 23.4 to 30 for no anxiety, any score greater than 30 for anxiety.

SECONDARY OUTCOMES:
emergence agitation difference between groups | postoperative every 5 minutes during 20 minutes
  Emergence agitation will be evaluated by PAED scale (pediatric anesthesia emergence delirium). The PAED scale involves five items: eye contact, purposeful actions, awareness of the surroundings, restlessness, inconsolability. First three items are scored as follows: 4= not at all, 3= just a little, 2= quite a bit, 1= very much, 0= extremely. Last two items are scored as follows: 0= not at all, 1= just a little, 2= quite a bit, 3= very much, 4= extremely. The scores of each item will summed to obtain a total score. PAED scale score of 10 or more will be defined as emergence delirium.
effect of parent's anxiety on child's anxiety | before premedication
  parent's anxiety will be evaluated by visual analog scale (VAS) at preoperative holding area

CONTACTS AND LOCATIONS:
Overall Officials: Ilkay Baran Akkuş, Principal Investigator — Diskapi Yildirim Beyazit Training Education Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training Research Hospital, Ankara, Altındag, Turkey (Türkiye)